CLINICAL TRIAL: NCT05414552
Title: Multicenter Retrospective Cohort Study on Patients Receiving Extracorporeal Photopheresis for Immune-related Adverse Events After Checkpoint Inhibitor Treatment
Brief Title: ECP for Immune-related Adverse Events After Checkpoint Inhibitor Treatment
Acronym: ECPforIRAE
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Professor, University of Freiburg
Other Study IDs: UKLFR06062022
Record Dates: First submitted 2022-06-06; First posted 2022-06-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Immune Related Adverse Events; Colitis; Hepatitis; Dermatitis
Keywords: extracorporeal photoperesis; immune modulation; immune checkpoint inhibitor
MeSH Terms: conditions — Colitis; Hepatitis; Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ECP treatment arm: ECP treatment per prtocol
  Interventions: Drug: ECP

INTERVENTIONS:
Drug: ECP — Treatment with ECP for irAEs with 2 cycles performed on two consecutive days, for the first 4 weeks repeated every week, and from week 5 to 12 repeated every two weeks

SUMMARY:
Preliminary data demonstrate that irAEs induced by immune checkpoint blockade can be successfully treated with ECP (Apostolova et al. NEJM 2020). Therefore this retrospective analysis is launched to validate the finding made with the individual patient in a larger patient cohort. The analysis will include the evaluation of safety of ECP treatment in patients with irAEs and collect data on the efficacy of ECP as a treatment for immune-related adverse events and its effect on tumor progression.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICI) have improved the long-term survival of patients with metastatic tumors. However, approximately 50% of the patients treated with ICI develop serious immune-related adverse events (irAE). A recent study reported that grade 3 or higher irAE occurred in 49 of 124 patients (39.5%) who received nivolumab/ipilimumab and in 41 of 123 patients (33.3%) who received nivolumab alone. Other studies report an overall frequency of grade 3-5 irAE in 24% - 59% of patients treated with nivolumab 1 mg/kg body weight and ipilimumab 3 mg/kg body weight. An incidence of 33.3% was reported when patients were treated with nivolumab 3 mg/kg body weight and ipilimumab 1 mg/kg body weight. The most common events reported during combined ICI treatment are diarrhea, rash, pruritus, hepatitis, hypothyroidism, neurological disease and pneumonitis. These numbers show that irAE are a particularly frequent complication of ICI and limit their use.

This retrospective analysis is launched to validate the finding made with the individual patient in a larger patient cohort. The analysis will include the evaluation of safety of ECP treatment in patients with irAEs and collect data on the efficacy of ECP as a treatment for immune-related adverse events and its effect on tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years
2. Written informed consent:

   * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines.
   * Subjects must be able to understand and willing to comply with scheduled visits, treatment schedule, laboratory tests and mandatory collection of blood, and other requirements of the study.
   * Subject Re-enrollment: This trial permits the re-enrollment of a subject that has discontinued the study as a screening failure. If re-enrolled, the subject must be re-consented.
3. Target population

   * Patients who have received treatment with an anti-PD-1, anti-PD-L1 or an anti-CTLA-4 antibody or any combination of these for any type of malignancy in the last 24 months before screening.
   * Patients should have clinical and/or histological evidence of immune-related adverse events as follows:

     * Colitis Diarrhea with increase of ≥4 stools over baseline No improvement after 72h treatment with at least 1 mg/kg BW/day prednisolone equivalent
     * Hepatitis Alanine aminotransferase and/or aspartate aminotransferase ≥3x ULN if baseline was normal; or ≥3x baseline if baseline was abnormal No improvement after 72h treatment with at least 1 mg/kg BW/day prednisolone equivalent
     * Pneumonitis Radiographic changes and new symptoms such as cough, dyspnea or chest pain No improvement after 72h treatment with 1 mg/kg BW/day prednisolone equivalent Dermatitis Skin erythema, maculopapular or pustulopapular rash covering ≥30% of the body surface area No improvement after 72h treatment with at least 1 mg/kg BW/day prednisolone equivalent
4. Maximum of one additional (second line) therapy after Steroid treatment before ECP starts (e.g. infliximab for colitis)
5. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 1 week prior to the start of study drug.
6. Women must not be breastfeeding.
7. ECOG performance status 0, 1, or 2

Exclusion Criteria:

1. Active treatment in a clinical study of any investigational agent within 14 days prior day 0 or within 5 half-lives of the study treatment, whichever is greater.
2. Positive result for HIV.
3. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
4. Mechanical ventilation or patients who have resting O2 saturation <90% by pulse-oximetry.
5. Patients who require vasopressors, and/or have NYHA class III or IV heart failure.
6. Uncontrolled hypertension or ventricular arrhythmias.
7. Previous or concurrent malignancies within the last 3 years of enrollment other than the disease for which checkpoint-inhibitor blockade was applied. Exceptions are adequately treated basal or squamous cell skin cancer, or any other cancer from which the subject has been disease-free for more than 3 years.
8. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data
9. Known allergies, hypersensitivity, or intolerance of methoxypsoralen, excipients, or similar compounds, heparin or similar compounds
10. Aphakia
11. Female patients of child-bearing potential who are not willing to use highly effective methods of contraception during the trial and at least 5 months after the ECP procedure (see also 10.9)
12. Inability to tolerate extracorporeal volume loss
13. Previous splenectomy
14. Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had develped irAEs after ICI and were treated with ECP outside of a clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Safety - treatment-related adverse events (AEs) and severe adverse events (SAEs) | 12 months after end of ECP
  To evaluate the rate of treatment-related adverse events (AEs) and severe adverse events (SAEs) in patients treated with ECP for immune-checkpoint inhibitor-induced colitis, pneumonitis, hepatitis or dermatitis.

SECONDARY OUTCOMES:
objective response rate | After 6 weeks of ECP therapy
  objective response rate (ORR) to treatment after 6 weeks of ECP therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center - University of Freiburg Albert-Ludwigs-University Freiburg Department of Medicine I, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
All information and data of this retrospective analysis will be made avaible to the public.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be made available after publication ofthe manuscript and from then on infinitively.

REFERENCES:
- [Result] Apostolova P, Unger S, von Bubnoff D, Meiss F, Becher B, Zeiser R. Extracorporeal Photopheresis for Colitis Induced by Checkpoint-Inhibitor Therapy. N Engl J Med. 2020 Jan 16;382(3):294-296. doi: 10.1056/NEJMc1912274. No abstract available. PMID 31940706
- [Result] Zeiser R, Polverelli N, Ram R, Hashmi SK, Chakraverty R, Middeke JM, Musso M, Giebel S, Uzay A, Langmuir P, Hollaender N, Gowda M, Stefanelli T, Lee SJ, Teshima T, Locatelli F; REACH3 Investigators. Ruxolitinib for Glucocorticoid-Refractory Chronic Graft-versus-Host Disease. N Engl J Med. 2021 Jul 15;385(3):228-238. doi: 10.1056/NEJMoa2033122. PMID 34260836